CLINICAL TRIAL: NCT06904586
Title: Evaluation of Anthropometric and Ultrasonographic Measurements With Different Machine Learning Methods in Predicting Difficult Intubation: A Prospective Observational Study
Brief Title: Anthropometric and US-Guided Difficult Intubation Prediction With ML Models
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Gizem Demir Şenoğlu, Ass. Prof., Duzce University
Other Study IDs: 2022/65
Record Dates: First submitted 2024-12-09; First posted 2025-04-01 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Difficult Endotracheal Intubation; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — ultrasonographic measurement The distance between the skin-trachea, skin-epiglotte, skin-vocal cord anterior commissure, skin-hyoid bone and mentum-hyoid bone will be recorded via ultrasonography on the case while the neck is in neutral position and extension.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients between the ages of 18 and 20 who will receive general anesthesia: ASA I-III patients over the age of 18 who meet the inclusion criteria to undergo general anesthesia
  Interventions: Other: Thyromental distance; Other: Neck circumference; Other: Mouth opening distance; Other: Distance from jawbone to hyoid bone with neck in neutral position; Other: Distance from jawbone to hyoid bone with neck in extension; Other: Distance between skin and trachea; Other: Distance between skin and epiglottis; Other: Distance between skin and anterior commissure of vocal cord:; Other: Distance between skin and hyoid bone; Other: Maximum Tongue Thickness

INTERVENTIONS:
Other: Thyromental distance — Distance between the chin and thyroid cartilage with a tape measure when the patient is in a neutral position
Other: Neck circumference — Measurement of neck circumference with a tape measure when the patient is in a neutral position
Other: Mouth opening distance — Distance between the upper and lower teeth at the point where the mouth opening is maximum when the patient is in a neutral position.
Other: Distance from jawbone to hyoid bone with neck in neutral position — Distance from mentum to hyoid bone with neck in neutral position by ultrasonography
Other: Distance from jawbone to hyoid bone with neck in extension — Ultrasound measurement of distance from mentum to hyoid bone with neck in extension
Other: Distance between skin and trachea — Ultrasound measurement of distance between skin and trachea
Other: Distance between skin and epiglottis — Distance between skin and epiglottis measured by ultrasonography
Other: Distance between skin and anterior commissure of vocal cord: — Distance between skin and anterior commissure of vocal cord measured by ultrasonography
Other: Distance between skin and hyoid bone — Distance between skin and hyoid bone measured by ultrasonography
Other: Maximum Tongue Thickness — Measurement of Maximal Tongue Thickness by Ultrasonography

SUMMARY:
The assessment and management of difficult airway is of critical importance. Unsuccessful airway management leads to serious mortality and morbidity. From the beginning of the pre-anesthesia examination, 3% to 13% of patients who are considered suitable for routine airway management may be difficult to intubate. Airway assessment issues include risk assessment and airway examination (bedside and forward) to estimate the risk of difficult airway or aspiration. Airway examination aims to determine the presence of upper airway pathologies or anatomical anomalies. Some physical characteristics are associated with difficult airways and unsuccessful intubation. Examples of these are; limited neck movement, snoring, short sternomental distance, neck circumference thickness, etc. Physical characteristics can be measured with a meter or more detailed upper airway ultrasonographic measurements. In this study, researchers aimed to evaluate the anthropometric and ultrasonographic measurement values of patients who underwent preoperative airway assessment and to see the predictability of difficult intubation with artificial intelligence-supported decision support programs.

DETAILED DESCRIPTION:
Difficult intubation, particularly unpredictable difficult intubation, is a challenging scenario for every anesthesiologist. Patients who are initially assessed as suitable for routine airway management may present as difficult to intubate in 5% to 22% of cases. Accurate evaluation and management of difficult airways are crucial, as failure in airway management can lead to serious morbidity and mortality.

Airway assessment helps identify predictable difficult airways, but it does not exclude patients with normal clinical evaluations who may still experience unpredictable difficult intubation. The primary goal of airway examination is to detect upper airway pathologies or anatomical anomalies. Several physical characteristics are associated with difficult airways and failed intubation, including limited neck mobility, snoring, a short sternomental distance, and increased neck circumference.

Common airway assessment tools, such as the Mallampati classification and the upper lip bite test, require patient cooperation, which limits their applicability in sedated, trauma, or unresponsive patients. The Cormack-Lehane classification, used during direct laryngoscopy, is invasive and does not allow for pre-procedural preparation. In this context, non-invasive, bedside, rapid, and accessible ultrasonographic assessments and anthropometric measurements have gained importance in predicting difficult airways.

With technological advancements, decision-support systems and artificial intelligence (AI)-assisted applications are increasingly used to prevent adverse outcomes. Successful airway management is particularly critical in high-risk patients, where rapid decision-making is essential. Easily accessible, bedside, non-invasive ultrasonographic measurements, integrated with AI-based learning programs, have the potential to predict difficult intubation in advance. This enables early preparation, timely interventions, and the reduction of life-threatening risks.

In this study, researchers aimed to predict difficult intubation preoperatively using non-invasive anthropometric and ultrasonographic upper airway measurements, combined with AI-assisted decision-support programs, without requiring any invasive procedures.

Our hypothesis is that preoperative airway assessment through anthropometric and ultrasonographic measurements, supported by AI-based decision-support programs, can accurately predict difficult intubation and facilitate early preparation

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients who will undergo general anesthesia

Exclusion Criteria:

* Pregnant women
* Those with congenital and/or acquired facial deformities
* Patients who have previously undergone upper neck airway surgery
* Patients with head and neck tumors
* Patients who will undergo thyroidectomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who were undergoing elective surgery were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gizem DEMIR SENOGLU, Principal Investigator — Duzce University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients Between the Ages of 18 and 20 Who Will Receive General Anesthesia
Started | 329
Completed | 329
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Between the Ages of 18 and 20 Who Will Receive General Anesthesia
Number analyzed (Participants) | 329
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 317
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 139
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 329

OUTCOME MEASURES:

1. Primary Outcome: Support Vector Machine Algorithm Percentage of Accuracy in Predicted Difficult Intubations
Description: The dataset, labeled based on expert assessment of difficult intubation, was classified using eight widely accepted machine learning algorithms: logistic regression (LR) [6], support vector machine (SVM) [7], random forest (RF) [8], K-nearest neighbors (KNN) [9], Gaussian naive Bayes (GNB) [10], CatBoost [11], XGBoost [12], and decision tree (DT) [13]. From the original 30 parameters, the 15 most influential features were selected based on feature extraction methods and literature relevance. Preprocessing steps included handling missing values, with incomplete records excluded. The dataset was split into training (80%) and test (20%) sets. Models were trained on the training set, with hyperparameter tuning performed via 5-fold cross-validation to avoid overfitting. Final model performance was evaluated on the independent test set.
Time Frame: Taking ultrasonographic and anthropometric measurements of each patient took approximately 20 minutes. Machine learning estimates for each patient are approximately 1 min.
Measure: Number (95% Confidence Interval); unit: percentage of estimate
Arm/Group | Patients Between the Ages of 18 and 20 Who Will Receive General Anesthesia
Number analyzed (Participants) | 329
percentage of estimate
  support vector macine Accuracy | 89.39 [80 to 95]
  Logistic Regression Accuracy | 77.27 [70 to 95]
  Random Forest Accuracy | 87.88 [80 to 95]
  Decision Tree Accuracy | 80.30 [80 to 95]
  K-Nearest Neighbors Accuracy | 74.24 [70 to 95]
  Gaussian Naive Bayes Accuracy | 71.21 [70 to 95]
  CatBoost Accuracy | 83.33 [80 to 95]
  XGBoost Accuracy | 81.82 [80 to 95]

ADVERSE EVENTS:
Time Frame: the time from preoperative preparation to delivery to surgery, 1 hour.
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored, but none observed.
Arm/Group | Patients Between the Ages of 18 and 20 Who Will Receive General Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/329
Serious Adverse Events (participants affected / at risk) | 0/329
Other Adverse Events (participants affected / at risk) | 0/329

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT06904586/Prot_SAP_ICF_000.pdf